CLINICAL TRIAL: NCT01683448
Title: The Effect of Perioperative Medications on the Outcomes of Patients Undergoing Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 298807
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Cardiac Diseases
Keywords: Perioperative medications; cardiac surgery; outcomes
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will be a retrospective study. The patient data from the electronic medical records and existing database will be collected and analyzed. Primary endpoints will be postoperative mortality (within 30 days) and overall complications and length of hospital stay. The secondary endpoints will be myocardial infarction, cardiac death, CHF, arrhythmia, ischemia, stroke, neurological complications, length of ICU stay, re-admission rate, infections, pulmonary complications, length of intubation time, length of ventilation time, and acute renal failure.

DETAILED DESCRIPTION:
Each year about 694,000 Americans have open-heart surgery including valve repairs, valve replacements, heart transplants, and coronary artery bypass graft (CABG) surgery [1]. The reported incidence of perioperative complications in these cardiac surgery patients is 4.5% while the prevalence varied from1.6% to 14.1% [2,3]. As the population ages, increased numbers of elderly patients with more advanced cardiac diseases and comorbidities are being referred for cardiac surgery. For these patients, postoperative cardiovascular complications (cardiac death, myocardial infarction (MI), ischemia, congestive heart failure (CHF), arrhythmia, stroke, and acute renal failure (ARF)) represent the major postoperative complications [4-6]. These complications translate into increased mortality, prolonged hospital stay and estimated costs exceeding $20 billion annually [7].

These events may be triggered by surgical stress responses that result in increased plasma levels of norepinephrine and epinephrine [8], myocardial oxygen supply demand imbalance, and plaque rupture [9].

Beta-blockers, ACE inhibitors, alfa2-agonists, Aspirin, statins, nitrates, anti-platelet medications and anticoagulation medications have been widely used in patients with coronary artery disease, hypertension and other heart diseases. Beta-blockers, ACE inhibitors and Aspirin statins have also been shown to have a positive impact on the outcomes of surgical and non-surgical treatments [10-11]. However, there are other studies which were unable to demonstrate the positive results of these medications on post-operative outcomes.

Based on the previous studies referenced above, we propose that the use of perioperative medications (Betablockers, ACE inhibitors, alfa2-agonists, Aspirin, statins, nitrates, anti-platelet medications, and anticoagulation medications) may provide cardiac protection for cardiac surgical patients. The specific aim of this study is to retrospectively investigate whether perioperative medication use is associated with decreases in the incidence of postoperative cardiovascular complications in patients undergoing elective cardiac surgery.

This study will be a retrospective study. The patient data from the electronic medical records and existing database will be collected and analyzed. Primary endpoints will be postoperative mortality (within 30 days) and overall complications and length of hospital stay. The secondary endpoints will be myocardial infarction, cardiac death, CHF, arrhythmia, ischemia, stroke, neurological complications, length of ICU stay, re-admission rate, infections, pulmonary complications, length of intubation time, length of ventilation time, and acute renal failure.

ELIGIBILITY:
Inclusion Criteria:

* All cardiac surgical patients

Exclusion Criteria:

* Non cardiac surgery

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiac surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
hemodynamic changes | In hospital
  blood pressure and heart rare

CONTACTS AND LOCATIONS:
Overall Officials: Hong Liu, M.D., Principal Investigator — UC Davis, Department of Anesthesiology and Pain Medicine
Locations (1):
- UC Davis, Medical Center, Sacramento, California, United States

REFERENCES:
- [Derived] Cheng H, Li Z, Young N, Boyd D, Atkins Z, Ji F, Liu H. The Effect of Dexmedetomidine on Outcomes of Cardiac Surgery in Elderly Patients. J Cardiothorac Vasc Anesth. 2016 Dec;30(6):1502-1508. doi: 10.1053/j.jvca.2016.02.026. Epub 2016 Mar 3. PMID 27435836
- [Derived] Ji F, Li Z, Nguyen H, Young N, Shi P, Fleming N, Liu H. Perioperative dexmedetomidine improves outcomes of cardiac surgery. Circulation. 2013 Apr 16;127(15):1576-84. doi: 10.1161/CIRCULATIONAHA.112.000936. Epub 2013 Mar 19. PMID 23513068